CLINICAL TRIAL: NCT03385668
Title: A Pilot Study to Evaluate the Efficacy and Safety of Pirfenidone in Patients With Pulmonary Fibrosis With Anti-myeloperoxydase (MPO) Antibodies or With Anti-MPO Associated Vasculitis."
Brief Title: Pilot Study of Pirfenidone in Pulmonary Fibrosis With Anti-myeloperoxydase Antibodies
Acronym: PIRFENIVAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Roche Pharma AG (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P161001J; 2017-002782-22 (EudraCT Number)
Record Dates: First submitted 2017-12-07; First posted 2017-12-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Fibrosis
Keywords: Pulmonary fibrosis; Antibodies, Antineutrophil Cytoplasmic; Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis; Pirfenidone; Microscopic Polyangiitis; Interstitial lung disease
MeSH Terms: conditions — Pulmonary Fibrosis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis; Lung Diseases, Interstitial | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pirfenidone (Experimental): All patients will receive Pirfenidone
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone at a dose of 2403 mg/day for 50 weeks, after a 2 weeks period of titration (801 mg/day for one week then 1602 mg/day for one week).

SUMMARY:
The purpose of this study is to determine wether pirfenidone is safe and effective in the treatment of pulmonary fibrosis with anti-myeloperoxydase (MPO) antibodies or pulmonary fibrosis with anti-MPO associated vasculitis.

DETAILED DESCRIPTION:
Pulmonary fibrosis can be associated with Anti-Neutrophil Cytoplasmic Antibody (ANCA) directed against MPO or with anti-MPO associated vasculitis, leading to increased disability and poor prognosis. The pathophysiology of this association remains unclear. Conventional therapies used for the treatment of vasculitis manifestations are often disappointing for the treatment of pulmonary fibrosis. The main cause of death in patients with anti-MPO ANCA associated vasculitis and associated pulmonary fibrosis is the progression of pulmonary fibrosis. No treatment has demonstrated efficacy to stabilize or improve pulmonary fibrosis associated with anti-MPO associated vasculitis.

Previous studies showed that Pirfenidone improves survival and pulmonary function in patients with idiopathic pulmonary fibrosis (IPF) and that Pirfenidone treatment is safe and well tolerated in IPF. Patients with anti-MPO associated vasculitis (or anti-MPO antibodies without vasculitis) and associated pulmonary fibrosis might benefit from the use of Pirfenidone. However, the efficacy and safety of pirfenidone in patients with anti-MPO associated vasculitis and associated pulmonary fibrosis has not been evaluated. This study was designed to assess the efficacy and safety of pirfenidone in patients with pulmonary fibrosis and anti-MPO ANCA associated vasculitis or anti-MPO antibodies without vasculitis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Presence of anti-MPO antibody (ELISA) at inclusion or during pulmonary fibrosis follow-up and/or diagnosis of anti-MPO associated vasculitis according to the 2012 Revised International Chapel Hill Consensus Conference definitions
* Definite or possible Usual Interstitial Pneumonia or Non Specific Interstitial Pneumonia based on high-resolution computed tomography
* Presence of pulmonary fibrosis, defined as a range of 50 to 90% of the %FVC and a range of 30 to 90% of the %DLCO
* Pulmonary fibrosis refractory (according to the investigator's judgment) to a conventional regimen used for anti-MPO associated vasculitis when a treatment against vasculitis has been used
* Have the ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information) and comply with the study protocol procedures (including required study visits)
* Have affiliation with a mode of social security (profit our being entitled).

Exclusion Criteria:

* Other type of systemic vasculitis;
* Active vasculitis defined by Birmingham Vasculitis Activity Score >3 (BVAS) ;
* Contraindication to Pirfenidone;
* Unable to perform pulmonary function test (PFT);
* Pregnancy or lactation. Women of childbearing capacity are required to have a negative serum pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using an effective method of birth control from the date of consent through the end of the study : implants of levonorgestrel; injectable progesterone; any intrauterine device (IUD) with a documented failure rate of less than 1% per year; oral contraceptives (either combined or progesterone only); double barrier method (condom, cervical cap or diaphragm with spermicidal agent); transdermal contraceptive patch; male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for the female subject;
* Any of the following liver function test criteria above specified limits: total bilirubin above 1,5 times the upper limit of normal (ULN), excluding patients with Gilbert's syndrome; aspartate (AST)/Glutamate Oxaloacétique Transaminase (SGOT) or alanine aminotransferase (ALT)/Glutamate Pyruvate Transaminase (SGPT), (AST/SGOT or ALT/SGPT) >3 × ULN; alkaline phosphatase >2.5 × ULN;
* Creatinine clearance (CrCl<30) mL/min, calculated using the Cockcroft-Gault formula at screening
* Current treatment with Nintedanib or past treatment with Nintedanib in the last 12 months;
* Current treatment with Fluvoxamine or past treatment with Fluvoxamine in the last 28 days before screening
* Prior use of Pirfenidone or known hypersensitivity to any of the components of study treatment;
* Expected to receive a lung transplant within 1 year from randomization or, on a lung transplant waiting list at randomization;
* Associated connective tissue disease (such as systemic sclerosis).;
* Electrocardiogram (ECG), with a heart-rate-corrected QT interval (corrected using Fridericia's formula, QTcF) ≥ 500 ms at Screening, or a family or personal history of long QT syndrome;
* Treatment with Cyclophosphamide in the last 3 months;
* Current smoking or past smoking in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy measured by the absolute change in percent predicted forced vital capacity (%FVC) | 52 weeks
  Treatment efficacy at Week 52 measured by the absolute change from baseline to Week 52 in percent predicted forced vital capacity (%FVC) :
  * Patients with progressive disease will be defined as absolute decline of 10% or more in %FVC. Missing values or death will be also considered as progressive.
  * Patients with non-progressive disease will be defined as improvement or no decline in %FVC or a decline of %FVC<10%.

SECONDARY OUTCOMES:
Adverse Events (AE) | 56 weeks corresponding to 28 days after the last dose of study drug
  Safety parameters reported in the period from baseline to 28 days after the last dose of the study drug:
  * Treatment-emergent AEs
  * Treatment-emergent Serious Adverse Events (SAE)
  * Treatment emergent Adverse Event of Special Interest (AESI)
  * Treatment-emergent treatment-related AEs
  * Treatment-emergent treatment-related SAEs
  * Treatment emergent related AESIs
  * AEs leading to early discontinuation of study treatment
  * Treatment-emergent deaths
  * Cause of death
  * Treatment-emergent changes in clinical laboratory findings
  * Vital signs
Treatment efficacy measured by the absolute change in percent predicted forced vital capacity (%FVC) | 24 weeks
  Treatment efficacy at Week 24 measured by the absolute change from baseline to Week 24 in percent predicted forced vital capacity (%FVC) :
  * Patients with progressive disease will be defined as absolute decline of 10% or more in %FVC. Missing values or death will be also considered as progressive.
  * Patients with non-progressive disease will be defined as improvement or no decline in %FVC or a decline of %FVC<10%.
Relative change in in percent predicted forced vital capacity | 52 weeks
  Relative change from baseline to Week 52 in percent predicted forced vital capacity (%FVC)
Absolute change in in percent predicted forced vital capacity | 52 weeks
  Relative and absolute change from baseline to Week 52 in percent predicted forced vital capacity (%FVC)
Relative change in in percent predicted forced vital capacity | 24 weeks
  Relative and absolute change from baseline to Week 24 in percent predicted forced vital capacity (%FVC)
Absolute change in in percent predicted forced vital capacity | 24 weeks
  Relative and absolute change from baseline to Week 24 in percent predicted forced vital capacity (%FVC)
Six minute walk test (6MWT) distance | 52 weeks
  Change from Baseline to Week 52 in the six minute walk test (6MWT) distance
Six minute walk test (6MWT) distance | 24 weeks
  Change from Baseline to Week 24 in the six minute walk test (6MWT) distance
Carbon Monoxide Diffusing Capacity (%DLCO) | 52 weeks
  Change from Baseline to Week 52 in the percent predicted Carbon Monoxide Diffusing Capacity (%DLCO)
Carbon Monoxide Diffusing Capacity (%DLCO) | 24 weeks
  Change from Baseline to Week 24 in the percent predicted Carbon Monoxide Diffusing Capacity (%DLCO)
Progression-free survival | 52 weeks
  Progression-free survival defined as the time to the first occurrence of any one of the following: a confirmed decrease of 10 percentage points or more in %FVC, a confirmed decrease of 15 percentage points or more in %DLCO, or death.
Dyspnea | 52 weeks
  Change from Baseline to Week 52 in dyspnea as measured by the New York Heart Association classification, the modified Borg scale and by the Saint-George's Respiratory Questionnaire (SGRQ).
Chest CT-scan | 52 weeks
  Change in Chest-CT scan abnormalities at Week 52 (evaluated after a centralized blinded review of the chest CT-scans).
Quality of Life assessed by the Health Assessment Questionnaire (HAQ) | 52 weeks
Quality of Life assessed by the Short Form-36 (SF-36) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan London, MD, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hervier B, Pagnoux C, Agard C, Haroche J, Amoura Z, Guillevin L, Hamidou MA; French Vasculitis Study Group. Pulmonary fibrosis associated with ANCA-positive vasculitides. Retrospective study of 12 cases and review of the literature. Ann Rheum Dis. 2009 Mar;68(3):404-7. doi: 10.1136/ard.2008.096131. Epub 2008 Oct 28. PMID 18957485
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312
- [Background] Lancaster L, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, King TE Jr, Lederer DJ, Lin Z, Nathan SD, Pereira CA, Swigris JJ, Valeyre D, Noble PW. Safety of pirfenidone in patients with idiopathic pulmonary fibrosis: integrated analysis of cumulative data from 5 clinical trials. BMJ Open Respir Res. 2016 Jan 12;3(1):e000105. doi: 10.1136/bmjresp-2015-000105. eCollection 2016. PMID 26835133